26.02.2025

Title: Methyl Alcohol Intoxication as a Public Health Issue: A 3-Year Retrospective Analysis

Yeliz Bilir\*, Banu Çevik\*, Akın Bilir\*, Elif Bombacı\*.

\*Department of Intensive Care, Kartal Dr Lütfi Kırdar City Hospital, İstanbul, Turkey

\*Corresponding author: Yeliz Bilir, M.D.

E-mail: dryelizbilir@yahoo.com

Address: Kartal Dr. Lütfi Kırdar City Hospital, D-100 Güney Yanyol No:47 Cevizli Mevkii

34865 Kartal / İSTANBUL

Phone: +90 5326657976

**Number of Tables: 5** 

**Number of Figures: 2** 

Word count: 2500

NCT Number: Not Available

Keywords: Methanol, Intoxication, Treatment, Outcomes.

#### STUDY PROTOCOL

The protocol must include the following items and necessary explanations:

#### 1. Title of the Study

"A Public Health Threat: Periodic Evaluation of Methanol Intoxication; A Retrospective Single-Center Study"

### 2. Study Center

Kartal Dr. Lütfi Kırdar City Hospital

#### 3. Principal Investigator

Assoc. Prof. Dr. Yeliz Bilir, Lütfi Kırdar City Hospital, Intensive Care Unit

### 4. Co-Investigators

- o Specialist Dr. Akın Bilir, Lütfi Kırdar City Hospital, Intensive Care Specialist
- o Prof. Dr. Banu Çevik, Lütfi Kırdar City Hospital, Anesthesiology and Reanimation
- Assistant Prof. Dr. Elif Bombacı, Lütfi Kırdar City Hospital, Intensive Care Unit

### 5. Rationale, Aim, and Importance of the Study

The aim of this study is to analyze and compare the cases of methanol poisoning admitted to our hospital, which is a major center in Istanbul, over the years in terms of frequency, patient profile, treatment methods, and survival rates.

**Secondary Objective:** To highlight the intensive care follow-up and treatment of this patient profile and provide a practical approach.

Patients diagnosed with methanol intoxication due to the consumption of counterfeit alcoholic beverages and admitted to the intensive care unit between 2022-2025 will be screened. These patients will be categorized into five-year periods based on their admission dates and compared in terms of demographic data, clinical characteristics, and survival outcomes.

#### 6. Type, Scope, and Design of the Planned Study

The study is designed as a retrospective cohort study.

### 7. Number and Characteristics of Patients to Be Included

All patients diagnosed with methanol intoxication due to the consumption of counterfeit alcoholic beverages and admitted to the intensive care unit between January 1, 2022, and March 1, 2025, will be included in the study, regardless of gender.

## 8. Parameters to Be Evaluated (Clearly Listed Individually)

The following parameters will be recorded:

- o Age, gender, and comorbidities of the patients
- o Glasgow Coma Scale (GCS) at admission and during follow-up
- Need for advanced life support (mechanical ventilation, vasopressor infusion, renal replacement therapy)
- APACHE-II, SOFA, and SAPS scores

- Blood gas values, routine biochemical values, troponin levels, GGT levels, urine output
- o Ethanol therapy, methanol levels, ethanol levels
- o Type of ingested substance (counterfeit alcohol or others)
- Presence of visual symptoms
- o Time of admission to intensive care after the incident
- o Length of stay in intensive care and hospital
- Survival status

## 9. Location and Personnel Responsible for Data Collection

The parameters included in the study will be collected by the researchers at the designated hospital.

## 10. Routine vs. Research-Specific Parameters

The data used in the study are part of routine intensive care treatments and do not incur additional costs.

# 11. Projected Study Duration, Start, and End Dates

The study will commence immediately after receiving Ethics Committee approval and is expected to be completed within six months.